CLINICAL TRIAL: NCT02705625
Title: A Randomised, Double-blind Placebo-controlled Phase IIa Study to Evaluate Efficacy, Safety and Tolerability of MIV-711 in Knee Joint Osteoarthritis
Brief Title: A Study to Evaluate the Efficacy, Safety and Tolerability of MIV-711 in Osteoarthritis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medivir (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MIV-711-201
Record Dates: First submitted 2016-03-07; First posted 2016-03-10 (Estimated); Results first posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-03

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — MIV-711

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MIV-711:1 (Experimental): MIV-711 for a total of 26 w
  Interventions: Drug: MIV-711
- MIV-711:2 (Experimental): MIV-711 for a total of 26 w
  Interventions: Drug: MIV-711
- Placebo (Placebo Comparator): Placebo for a total of 26 w
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MIV-711 — MIV-711 administered orally once daily
  Arms: MIV-711:1; MIV-711:2
Drug: Placebo — Placebo manufactured to mimic MIV-711 capsule.
  Arms: Placebo

SUMMARY:
This is a multicentre, randomised, placebo-controlled, double-blind, three-arm parallel, Phase IIa study to evaluate the efficacy, safety and tolerability of MIV-711 in patients with knee osteoarthritis (OA).

ELIGIBILITY:
Inclusion Criteria:

* Current average knee pain, defined as pain in either knee, within 1 week before visit 1, for which the patient gives a severity score of ≥4, <10 on a 0-10 NRS (Numeric Rating Scale).
* Inclusive of 40-80 years old.
* Diagnosis of primary knee osteoarthritis

Exclusion Criteria:

* The presence of any inflammatory arthritis
* Any generalized pain condition that may interfere with the evaluation of the target knee pain (e.g., fibromyalgia) as judged by the investigator.
* Any clinically severe or significant uncontrolled concurrent illness, which, in the opinion of the Investigator, would impair ability to give informed consent or take part in or complete this clinical study.
* Known or suspected intolerance or hypersensitivity to the investigational product, closely related compounds, or any of the stated ingredients.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2016-01-28 (Actual); Primary Completion 2017-05-23 (Actual); Study Completion 2017-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Conaghan, Professor, Principal Investigator — Leeds Institute of Rheumatic and Musculoskeletal Medicine
Locations (6):
- MC Comac Medical, Sofia, Bulgaria
- LCC ARENSIA Exploratory Medicine, Tbilisi, Georgia
- PAREXEL Berlin Early Phase Clinical Unit, Berlin, Germany
- LCC ARENSIA Exploratory Medicine, Chisinau, Moldova
- SC ARENSIA Exploratory Medicine SRL, Bucharest, Romania
- University of Leeds, Leeds Institute of Rheumatic and Musculoskeletal Medicine, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- MIV-711:100 mg: MIV-711 100 mg administered orally once daily for a total of 26 weeks
- MIV-711:200 mg: MIV-711 200 mg administered orally once daily for a total of 26 weeks
- Placebo: Placebo manufactured to mimic MIV-711 capsule administered orally once daily for a total of 26 weeks
Period: Overall Study
Arm/Group | MIV-711:100 mg | MIV-711:200 mg | Placebo
Started | 82 | 82 | 80
Completed | 74 | 72 | 69
Not Completed | 8 | 10 | 11
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Adverse Event | 6 | 5 | 2
Not completed — Death | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 4 | 5
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Non-compliance | 0 | 1 | 1
Not completed — Overdosing | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: mITT population used in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | MIV-711:100 mg | MIV-711:200 mg | Placebo | Total
Number analyzed (Participants) | 82 | 81 | 77 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (6.58) | 62.0 (7.33) | 62.3 (6.59) | 61.8 (6.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 58 | 62 | 184
  Male | 18 | 23 | 15 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 2
  White | 82 | 81 | 75 | 238
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Romania | 3 | 2 | 3 | 8
  United Kingdom | 0 | 1 | 1 | 2
  Moldova | 26 | 29 | 36 | 91
  Georgia | 13 | 13 | 7 | 33
  Bulgaria | 14 | 14 | 9 | 37
  Germany | 26 | 22 | 21 | 69

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Scale (NRS) Average Target Knee Pain Score at Week 26
Description: Change from Visit 2 (Baseline) to Visit 8 (Week 26) in NRS average target knee pain score.
  NRS (Numeric rating scale) ranges from 0 indicating -"no pain", to 10 indicating - "pain as bad as it could be".
Time Frame: baseline and 26 weeks
Population: As there were discontinuations in the study, not all patients in the mITT population had an assessment at week 26. The analysis population is therefore equal to the number of patients completing the study for this outcome measure.
Measure: Mean (Standard Deviation); unit: score
Groups:
- Placebo: Placebo, manufactured to mimic MIV-711 capsule, administered orally once daily for a total of 26 weeks
Arm/Group | MIV-711:100 mg | MIV-711:200 mg | Placebo
Number analyzed (Participants) | 74 | 72 | 69
score | -1.7 (2.01) | -1.5 (1.95) | -1.3 (2.15)
Statistical Analysis 1: Comparison: MIV-711:200 mg vs Placebo; A linear mixed model based on the mITT population was used. The model included fixed factors for treatment, time (measured in weeks), the interaction for treatment by time, baseline analgesic user (Yes/No), and random effect for clinical site. Baseline NRS was included as a covariate for adjustment. An unstructured covariance matrix was used to model the covariance pattern in the mixed effects model; Test type: Superiority — For the primary endpoint, the Type I error for the tests of the two doses was protected by performing a fixed-sequence multiple-testing procedure in the following order: Step 1: 200 mg versus placebo Step 2: 100 mg versus placebo The second step was only considered as confirmatory provided the previous step was significant at a one-sided 5%-level (p<0.05). If the previous step was not significant, the analysis of the following step was considered descriptive; p = 0.4055, Mixed Models Analysis — The p-values reported is from Step 1 (comparing 200 mg versus placebo). The corresponding p-value from Step 2 (comparing 100 mg versus placebo) was 0.1458; Mean Difference (Final Values) = -0.0761, 95% CI 2-sided [-0.703 to 0.55]

2. Secondary Outcome: Magnetic Resonance Imaging (MRI) Bone Area of the Target Knee at Week 26
Description: Change from Visit 2 (Baseline) to Visit 8 (Week 26) in MRI (Magnetic Resonance Imaging;) bone area of the target knee in mm^2.
Time Frame: baseline and 26 weeks
Population: As there were discontinuations in the study, not all patients in the mITT population had an MRI assessment at week 26. In addition, there were patients with non valid MRIs. The analysis population is therefore smaller than the Participant Flow.
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | MIV-711:100 mg | MIV-711:200 mg | Placebo
Number analyzed (Participants) | 69 | 69 | 66
mm^2 | 8.1290 (31.10846) | 8.2142 (29.39941) | 23.2234 (32.68365)
Statistical Analysis 1: Comparison: MIV-711:200 mg vs Placebo; A linear mixed model based on the mITT population was used. The model included fixed factors for treatment, time (measured in weeks), the interaction for treatment-by-time, baseline analgesic user (Yes/No), and random effect for clinical site. Baseline knee joint MRI bone area was included as a covariate for adjustment. An unstructured covariance matrix was used to model the covariance pattern in the mixed effects model; Test type: Superiority — One model is fit for all comparison groups (MIV-711 200 mg, MIV-711 100 mg and placebo). This analysis reports the contrast that compares 200 mg versus placebo with respect to mean change from baseline in knee joint MRI bone area at Week 26; p = 0.0036, Mixed Models Analysis — p-values reported are unadjusted p-values for tests of significance for the upper one-tailed alternative hypothesis Ha: bone area increase is lower in the active treatment arm compared to placebo; Mean Difference (Final Values) = -14.7, 95% CI 2-sided [-25.3 to -4.02]
Statistical Analysis 2: Comparison: MIV-711:100 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — One model is fit for all comparison groups (MIV-711 200 mg, MIV-711 100 mg and placebo). This analysis reports the contrast that compares 100 mg versus placebo with respect to mean change from baseline in knee joint MRI bone area at Week 26; p = 0.0023, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -15.4, 95% CI 2-sided [-26 to -4.83]

3. Secondary Outcome: Magnetic Resonance Imaging (MRI) of Cartilage Thickness (Femur) at Week 26
Description: Change from Visit 2 (baseline) to Visit 8 (week 26) in MRI cartilage thickness in the Central Medial Femur Region of the target knee in mm.
Time Frame: baseline and 26 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | MIV-711:100 mg | MIV-711:200 mg | Placebo
Number analyzed (Participants) | 69 | 69 | 66
mm | 0.0077 (0.19258) | -0.0171 (0.24113) | -0.0658 (0.21904)
Statistical Analysis 1: Comparison: MIV-711:200 mg vs Placebo; A linear mixed model based on the mITT population was used. The model included fixed factors for treatment, time (measured in weeks), the interaction for treatment-by-time, baseline analgesic user (Yes/No), and random effect for clinical site. Baseline MRI of cartilage thickness was included as a covariate for adjustment. An unstructured covariance matrix was used to model the covariance pattern in the mixed effects model; Test type: Superiority — One model is fit for all comparison groups (MIV-711 200 mg, MIV-711 100 mg and placebo). This analysis reports the contrast that compares 200 mg versus placebo with respect to mean change from baseline in MRI of cartilage thickness (Femur Region) at Week 26; p = 0.1253, Mixed Models Analysis — p-values reported are unadjusted p-values for tests of significance for the upper one-tailed alternative hypothesis Ha: MRI of cartilage thinning (Femur Region) is lower in the active treatment arm compared to placebo; Mean Difference (Final Values) = 0.0436, 95% CI 2-sided [-0.031 to 0.118]
Statistical Analysis 2: Comparison: MIV-711:100 mg vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority — One model is fit for all comparison groups (MIV-711 200 mg, MIV-711 100 mg and placebo). This analysis reports the contrast that compares 100 mg versus placebo with respect to mean change from baseline in MRI of cartilage thickness (Femur Region) at Week 26; p = 0.0225, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.0761, 95% CI 2-sided [0.00173 to 0.15]

4. Secondary Outcome: Normalised Western Ontario & McMaster Universities Osteoarthritis Index (WOMAC) Pain Score
Description: Change from Visit 2 (Baseline) to Visit 8 (Week 26) in normalised WOMAC pain score. The WOMAC responses are scored using an 11-point NRS where 0=none and 10=extreme. There are 5 questions in the WOMAC pain scale which is summed up for the total WOMAC score, leading to a range of 0 to 50. The total WOMAC pain score has been standardised to a scale with a range from 0 to 100 (where 100 is extreme pain):
  - Normalised WOMAC pain score = Total WOMAC pain score multiplicated with 2.
Time Frame: baseline and 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | MIV-711:100 mg | MIV-711:200 mg | Placebo
Number analyzed (Participants) | 74 | 72 | 69
score | -16.6 (19.35) | -13.0 (18.6) | -9.8 (21.89)
Statistical Analysis 1: Comparison: MIV-711:200 mg vs Placebo; A linear mixed model based on the mITT population was used. The model included fixed factors for treatment, time (measured in weeks), the interaction for treatment-by-time,baseline analgesic user (Yes/No), and random effect for clinical site. Baseline WOMAC Pain score was included as a covariate for adjustment. An unstructured covariance matrix was used to model the covariance pattern in the mixed effects model; Test type: Superiority — One model is fit for all comparison groups (MIV-711 200 mg, MIV-711 100 mg and placebo). This analysis reports the contrast that compares 200 mg versus placebo with respect to mean change from baseline in WOMAC Pain score at Week 26; p = 0.2887, Mixed Models Analysis — p-values reported are unadjusted p-values for tests of significance for the lower one-tailed alternative hypothesis Ha: Reduction in WOMAC Pain score is higher in the active treatment arm compared to placebo; Mean Difference (Final Values) = -1.77, 95% CI 2-sided [-8.02 to 4.48]
Statistical Analysis 2: Comparison: MIV-711:100 mg vs Placebo; A linear mixed model based on the mITT population was used. The model included fixed factors for treatment, time (measured in weeks), the interaction for treatment-by-time, baseline analgesic (Yes/No) and random effect for clinical site. Baseline WOMAC Pain score was included as a covariate for adjustment. An unstructured covariance matrix was used to model the covariance pattern in the mixed effects model; Test type: Superiority — One model is fit for all comparison groups (MIV-711 200 mg, MIV-711 100 mg and placebo). This analysis reports the contrast that compares 100 mg versus placebo with respect to mean change from baseline in WOMAC Pain score at Week 26; p = 0.0753, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]; Mean Difference (Final Values) = -4.55, 95% CI 2-sided [-10.8 to 1.67]

5. Secondary Outcome: Normalised Western Ontario & McMaster Universities Osteoarthritis Index (WOMAC) Difficulty Score
Description: Change from Visit 2 (Baseline) to Visit 8 (Week 26) in normalised WOMAC difficulty score. The WOMAC responses are scored using an 11-point NRS where 0=none and 10=extreme. There are 17 questions in the WOMAC difficulty scale which is summed up for the total WOMAC difficulty score, leading to a range of 0 to 170. The total WOMAC difficulty score has been standardised to a scale with a range from 0 to 100 (where 100 is extreme pain):
  - Normalised WOMAC difficulty score = Total WOMAC difficulty score divided with 1.7
Time Frame: baseline and 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | MIV-711:100 mg | MIV-711:200 mg | Placebo
Number analyzed (Participants) | 74 | 72 | 69
score | -16.39 (20.937) | -13.95 (20.668) | -9.9 (21.862)
Statistical Analysis 1: Comparison: MIV-711:200 mg vs Placebo; A linear mixed model based on the mITT population was used. The model included fixed factors for treatment, time (measured in weeks), the interaction for treatment-by-time, baseline analgesic (Yes/No) and random effect for clinical site. Baseline WOMAC Difficulty score was included as a covariate for adjustment. An unstructured covariance matrix was used to model the covariance pattern in the mixed effects model; Test type: Superiority — One model is fit for all comparison groups (MIV-711 200 mg, MIV-711 100 mg and placebo). This analysis reports the contrast that compares 200 mg versus placebo with respect to mean change from baseline in WOMAC difficulty score at Week 26; p = 0.2898, Mixed Models Analysis — p-values reported are unadjusted p-values for tests of significance for the lower one-tailed alternative hypothesis Ha: Reduction in WOMAC Difficulty score is higher in the active treatment arm compared to placebo; Mean Difference (Final Values) = -1.84, 95% CI 2-sided [-8.38 to 4.7]
Statistical Analysis 2: Comparison: MIV-711:100 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority — One model is fit for all comparison groups (MIV-711 200 mg, MIV-711 100 mg and placebo). This analysis reports the contrast that compares 100 mg versus placebo with respect to mean change from baseline in WOMAC difficulty score at Week 26; p = 0.1262, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Final Values) = -3.78, 95% CI 2-sided [-10.3 to 2.72]

6. Secondary Outcome: Normalised Western Ontario & McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Score
Description: Change from Visit 2 (Baseline) to Visit 8 (Week 26) in normalised WOMAC stiffness score. The WOMAC responses are scored using an 11-point NRS where 0=none and 10=extreme. There are 2 questions in the WOMAC stiffness scale which is summed up for the total WOMAC stiffness score, leading to a range of 0 to 20. The total WOMAC stiffness score has been standardised to a scale with a range from 0 to 100 (where 100 is extreme pain):
  - Normalised WOMAC stiffness score = Total WOMAC stiffness score multiplicated with 5
Time Frame: baseline and 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score
Arm/Group | MIV-711:100 mg | MIV-711:200 mg | Placebo
Number analyzed (Participants) | 74 | 72 | 69
score | -17 (24.69) | -14.5 (22.71) | -9.8 (24.71)
Statistical Analysis 1: Comparison: MIV-711:200 mg vs Placebo; A linear mixed model based on the mITT population was used. The model included fixed factors for treatment, time (measured in weeks), the interaction for treatment-by-time, baseline analgesic (Yes/No) and random effect for clinical site. Baseline WOMAC Stiffness score was included as a covariate for adjustment. An unstructured covariance matrix was used to model the covariance pattern in the mixed effects model; Test type: Superiority — One model is fit for all comparison groups (MIV-711 200 mg, MIV-711 100 mg and placebo). This analysis reports the contrast that compares 200 mg versus placebo with respect to mean change from baseline in WOMAC stiffness score at Week 26; p = 0.2, Mixed Models Analysis — p-values reported are unadjusted p-values for tests of significance for the lower one-tailed alternative hypothesis Ha: Reduction in WOMAC Stiffness score is higher in the active treatment arm compared to placebo; Mean Difference (Final Values) = -3.07, 95% CI 2-sided [-10.2 to 4.1]
Statistical Analysis 2: Comparison: MIV-711:100 mg vs Placebo; A linear mixed model based on the mITT population was used. The model included fixed factors for treatment, time (measured in weeks), the interaction for treatment-by-time, baseline analgesic user (Yes/No), and random effect for clinical site. Baseline WOMAC stiffness score was included as a covariate for adjustment. An unstructured covariance matrix was used to model the covariance pattern in the mixed effects model; Test type: Superiority — One model is fit for all comparison groups (MIV-711 200 mg, MIV-711 100 mg and placebo). This analysis reports the contrast that compares 100 mg versus placebo with respect to mean change from baseline in WOMAC stiffness score at Week 26; p = 0.0861, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -4.95, 95% CI 2-sided [-12.1 to 2.17]

7. Secondary Outcome: Serum C-terminal Telopeptide of Collagen Type I (CTX-I) at Week 26
Description: Change from Visit 2 (baseline) to Visit 8 (week 26) in serum CTX-I, a biomarker for bone resorption.
Time Frame: baseline and 26 weeks
Population: As there were discontinuations in the study, not all patients in the mITT population had an assessment at week 26. In addition, there was one missing sample for serum CTX-I. The analysis population is therefore smaller than in the Participant Flow.
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | MIV-711:100 mg | MIV-711:200 mg | Placebo
Number analyzed (Participants) | 74 | 71 | 69
ug/L | -0.1209 (0.16733) | -0.2575 (0.19931) | 0.0000 (0.16165)
Statistical Analysis 1: Comparison: MIV-711:200 mg vs Placebo; A linear mixed model based on the mITT population was used. The model included fixed factors for treatment, time (measured in weeks), the interaction for treatment-by-time, baseline analgesic user (Yes/No), and random effect for clinical site. Baseline CTX-I score was included as a covariate for adjustment. An unstructured covariance matrix was used to model the covariance pattern in the mixed effects model; Test type: Superiority — One model is fit for all comparison groups (MIV-711 200 mg, MIV-711 100 mg and placebo). This analysis reports the contrast that compares 200 mg versus placebo with respect to mean change from baseline in CTX-I score at Week 26; p < 0.0001, Mixed Models Analysis — p-values reported are unadjusted p-values for tests of significance for the upper one-tailed alternative hypothesis Ha: CTX-I score is lower in the active treatment arm compared to placebo; Mean Difference (Final Values) = -0.254, 95% CI 2-sided [-0.302 to -0.206]
Statistical Analysis 2: Comparison: MIV-711:100 mg vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority — One model is fit for all comparison groups (MIV-711 200 mg, MIV-711 100 mg and placebo). This analysis reports the contrast that compares 100 mg versus placebo with respect to mean change from baseline in CTX-I score at Week 26; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 7, analysis 1]; Mean Difference (Final Values) = -0.145, 95% CI 2-sided [-0.193 to -0.0983]

8. Secondary Outcome: Creatinine Corrected Urine C-terminal Telopeptide of Collagen Type II (CTX-II) at Week 26
Description: Change from Visit 2 (baseline) to Visit 8 (week 26) in creatinine corrected urine CTX-II, a biomarker for cartilage degradation.
Time Frame: baseline and 26 weeks
Population: As there were discontinuations in the study, not all patients in the mITT population had an assessment at week 26. In addition, there was two missing samples for urine CTX-II. The analysis population is therefore smaller than in the Participant Flow.
Measure: Mean (Standard Deviation); unit: ng/mmol
Arm/Group | MIV-711:100 mg | MIV-711:200 mg | Placebo
Number analyzed (Participants) | 73 | 72 | 68
ng/mmol | -138.0 (198.68) | -242.5 (266.56) | 28.4 (225.69)
Statistical Analysis 1: Comparison: MIV-711:200 mg vs Placebo; A linear mixed model based on the mITT population was used. The model included fixed factors for treatment, time (measured in weeks), the interaction for treatment-by-time, baseline analgesic user (Yes/No), and random effect for clinical site. Baseline CTX-II score was included as a covariate for adjustment. An unstructured covariance matrix was used to model the covariance pattern in the mixed effects model; Test type: Superiority — One model is fit for all comparison groups (MIV-711 200 mg, MIV-711 100 mg and placebo). This analysis reports the contrast that compares 200 mg versus placebo with respect to mean change from baseline in CTX-II score at Week 26; p < 0.0001, Mixed Models Analysis — p-values reported are unadjusted p-values for tests of significance for the upper one-tailed alternative hypothesis Ha: CTX-II score is lower in the active treatment arm compared to placebo; Mean Difference (Final Values) = -270, 95% CI 2-sided [-339 to -201]
Statistical Analysis 2: Comparison: MIV-711:100 mg vs Placebo; A linear mixed model based on the mITT population was used. The model included fixed factors for treatment, time (measured in weeks), the interaction for treatment-by- time, baseline analgesic user (Yes/No), and random effect for clinical site. Baseline CTX-II score was included as a covariate for adjustment. An unstructured covariance matrix was used to model the covariance pattern in the mixed effects model; Test type: Superiority — One model is fit for all comparison groups (MIV-711 200 mg, MIV-711 100 mg and placebo). This analysis reports the contrast that compares 100 mg versus placebo with respect to mean change from baseline in CTX-II score at Week 26; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 8, analysis 1]; Mean Difference (Final Values) = -193, 95% CI 2-sided [-262 to -124]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from signing the Informed Consent Form to the Follow up visit (4 weeks after end of treatment).
Arm/Group | MIV-711:100 mg | MIV-711:200 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/82 | 1/80
Serious Adverse Events (participants affected / at risk) | 3/82 | 2/82 | 1/80
Other Adverse Events (participants affected / at risk) | 33/82 | 27/82 | 33/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MIV-711:100 mg (N=82) | MIV-711:200 mg (N=82) | Placebo (N=80)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Prinzmetal angina (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis chronic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MIV-711:100 mg (N=82) | MIV-711:200 mg (N=82) | Placebo (N=80)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 4 (4)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 4 (4)
Headache (Nervous system disorders) | 5 (6) | 5 (5) | 6 (8)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 (7) | 6 (6) | 7 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 2 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (7) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 8 (8) | 7 (9) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-07-20): https://cdn.clinicaltrials.gov/large-docs/25/NCT02705625/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-22): https://cdn.clinicaltrials.gov/large-docs/25/NCT02705625/SAP_001.pdf